CLINICAL TRIAL: NCT02158208
Title: Study of the T CD8 Immune Response in Horton's Disease
Acronym: Horton CD8
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: SAMSON APJ 2013
Record Dates: First submitted 2014-03-05; First posted 2014-06-06 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Horton's Disease
Keywords: before any treatment; at the diagnosis
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients with HD
  Interventions: Other: Blood sample drawn into a 5 mL dry tube at the diagnosis and after 3 months of treatment; Other: 16 blood samples drawn into 6 mL heparinized tubes at the diagnosis and after 3 months of treatment
- Controls
  Interventions: Other: Blood sample drawn into a 5 mL dry tube; Other: 16 blood samples drawn into 6 mL heparinized tubes

INTERVENTIONS:
Other: Blood sample drawn into a 5 mL dry tube at the diagnosis and after 3 months of treatment
  Groups: Patients with HD
Other: 16 blood samples drawn into 6 mL heparinized tubes at the diagnosis and after 3 months of treatment
  Groups: Patients with HD
Other: Blood sample drawn into a 5 mL dry tube
  Groups: Controls
Other: 16 blood samples drawn into 6 mL heparinized tubes
  Groups: Controls

SUMMARY:
The research hypothesis is that T lymphocytes CD8 play a role in the physiopathology of Horton's disease.

At the inclusion visit, patients will have, as is the case in the usual strategy:

* A complete clinical examination carried out by the doctor in charge of the patient
* ESR, and CRP and fibrinogen assay
* A full blood count for leukocytes and lymphocytes
* A biopsy of the temporal artery (TAB) to screen for signs of vascularitis, suggesting Horton's disease. The clinician in charge of the patient will decide if a second biopsy is necessary. The biopsy will be sent to and analysed at Anatomy and Pathological cytology service. Immunohistochemical analyses will be done if the TAB is positive.

In addition to the standard clinical examination and complementary examinations relative to the patients' pathology, the following will be done:

* Lymphocyte immunophenotyping for the quantity of T CD4 (cluster of differentiation 4) and CD8 lymphocytes, B lymphocytes and natural killer lymphocytes. This will make it possible to calculate the absolute value for different T lymphocyte populations.
* A blood sample drawn into a dry 5 mL tube (large yellow) to isolate the serum, which will be stored at -80°C for future assays for cytokines and other biomarkers of interest for Horton's disease.
* 16 blood samples drawn into 6 mL heparinized tubes (large green). These will be used immediately for cytometric and functional analyses.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Patients who have provided written informed consent
* Patients covered by national health insurance
* Age > 50 years
* Patients with Horton's disease at the diagnosis before any treatment

Horton's disease is defined by American College of Rheumatology criteria, the diagnosis is made if any 3 of the following 5 criteria are associated:

* age at the onset of the disease 50 years or above
* recent onset localised headache
* indurated temporal artery or decrease/absence of temporal pulse
* erythrocyte sedimentation rate (ESR) above 50 mm for the first hour (or CRP>20 mg/L)
* positive TAB showing vascularitis with infiltration of mononucleated cells or granulomatous inflammation with or without giant cells.

Controls Controls will be healthy volunteers recruited from blood donors of Dijon CHU, voluntary hospital personnel (nurses, doctors, laboratory technicians and secretaries) and patients without infectious or inflammatory disease, cancer or auto-immune disease (CRP<5mg/L) recruited in the department of the investigators at Dijon CHU. They will be matched for age and sex.

* Age > 50 years
* Patients covered by national health insurance
* who have provided written informed consent to take part
* Absence of inflammatory syndrome (CRP<5 mg /L)

Exclusion Criteria:

* Any patient not meeting inclusion criteria
* Patient treated with corticoids or immunosuppressants in the month preceding inclusion
* Patients treated with chemotherapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting Horton's disease at the diagnosis before any treatment
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-07-25 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
The percentage of cytotoxic T lymphocytes CD8 (CD8+perforin+granzyme B+) | Change from baselines the percentage of cytotoxic T lymphocytes CD8 at 3 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Derived] Maldiney T, Greigert H, Martin L, Benoit E, Creuzot-Garcher C, Gabrielle PH, Chassot JM, Boccara C, Balvay D, Tavitian B, Clement O, Audia S, Bonnotte B, Samson M. Full-field optical coherence tomography for the diagnosis of giant cell arteritis. PLoS One. 2020 Aug 31;15(8):e0234165. doi: 10.1371/journal.pone.0234165. eCollection 2020. PMID 32866179